CLINICAL TRIAL: NCT04093414
Title: Left Bundle Area Versus Selective His Bundle Pacing (LEFTBASH): Single Center, Open Label, Randomized Pilot Study to Evaluate Capture Thresholds and Acute Echocardiographic Hemodynamic Characteristics
Brief Title: Left Bundle Area Versus Selective His Bundle Pacing
Acronym: LEFTBASH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow enrollment
Sponsor: David Haines, MD (Other)
Responsible Party: Sponsor-Investigator, David Haines, MD, Director, Electrophysiology and Heart Rhythm Centre, Corewell Health East
Organization: Corewell Health East (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-191
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Results first posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-06

CONDITIONS: Bradycardia; Sinus Node Dysfunction; Atrioventricular Block
Keywords: Pacemaker; Bundle of His; Left Bundle Branch
MeSH Terms: conditions — Bradycardia; Sick Sinus Syndrome; Atrioventricular Block

STUDY DESIGN:
Intervention Model Description: Single center, open label, randomized, prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Selective or Non selective His Bundle Pacing (Active Comparator): Pacemaker wires placed in Bundle of His
  Interventions: Device: Select Secure pacing lead
- Left Bundle Area Pacing (Active Comparator): Pacemaker wires placed in Left Bundle Branch area
  Interventions: Device: Select Secure pacing lead

INTERVENTIONS:
Device: Select Secure pacing lead — A Select Secure pacing lead is placed in the bundle of His or Left bundle branch area based upon randomization
  Other Names: Select Secure 3830, 69 cm, Medtronic Inc.

SUMMARY:
This is a voluntary research study to find out which location in the heart a pacemaker wire is the most efficient for a patient's heart and for battery life. Patients who volunteer and are eligible for the study will be randomized to receive one of two positions for the wire to be screwed into, in addition to studying multiple positions in the heart during the pacemaker insertion. Enrolled patients will be in the study for 1 year. They will also have an Ultrasound of their heart performed to assess how the pacemaker wire is affecting their heart. Pacemakers are connected to the heart by wires that are screwed into the heart. The wires can be connected to the heart in different places, which can affect how well the heart beats over time. The typical position is at the tip of the heart. This position may cause the heart to beat inefficiently. Over time, this could lead to weakened heart muscle, irregular heart rhythm, and more hospitalizations. The heart has special muscle cells and fibers that carry electrical signals through and around the heart. An alternative spot to place the pacemaker wire is in an area where these special cells are grouped together (called the HIS bundle). The pacemaker wire can be connected to the heart at a location which may allow the heart to beat more efficiently when compared to putting the wire at traditional spots in the heart (called HIS bundle pacing). However, sometimes connecting the wire into the HIS bundle may cause the pacemaker battery to wear out faster. Physicians can also connect the pacemaker wired near the HIS bundle (called Left left Bundle bundle area pacing). The study physicians hope this will allow the heart to beat more efficiently without causing the battery to wear out faster. The study physicians would like to study how different wire positions change heart beat efficiency and how long the pacemaker battery lasts when the wires are placed in different locations. This study will connect the pacemaker wire at either the HIS Bundle or the left bundle area pacing, to see how effectively the heart pumps and how much battery is being used.

DETAILED DESCRIPTION:
This is a single center, open label, prospective randomized pilot study to evaluate the capture threshold of His Bundle versus left bundle area pacing. Secondary analysis will focus on changes in left ventricular performance and mechanical synchrony. Symptomatic bradyarrhythmias are effectively treated with cardiac pacemakers.The amount of pacing by the lead positioned in the bottom chamber of the heart at traditional sites such as the right ventricular apex have been associated with increased rates of atrial fibrillation, heart failure, and mortality. Traditional pacing sites result in cardiac electromechanical dyssynchrony, for which alternate pacing sites to minimize these untoward effects have been sought. HIS bundle pacing, which utilizes a patient's native conduction, has demonstrated improved electrical synchrony and left ventricular function when compared to traditional pacing at the tip of the bottom chamber. Barriers to wide spread application to this technique include the His bundle anatomic location and its attendant difficulties associated with implant, as well as higher capture thresholds leading to decreased battery duration of the pacemaker. An alternative to HIS bundle pacing is placing the lead just past the HIS bundle area, which is further in the heart, and to actively fixate the lead into the interventricular septum. This is referred to as Left Bundle Pacing, as it may electrically capture the left bundle, which would simulate a patient's native conduction. The researchers will evaluate the two different pacing sites (HIS bundle and Left Bundle area sites) to determine how effectively the heart pumps with each pacing site.

Patients requiring pacemaker implant will be screened for study eligibility and approached for informed consent. Baseline assessments including echocardiogram and ECG will be obtained. A standard of care echo done within 3 months of the procedure will be used as the baseline echo. Once enrolled, the researchers will randomize patients to one of two arms. One arm will fixate the ventricular pacemaker lead to the HIS bundle area while the other arm will have the leads fixed into the left bundle area. The pacemaker wires will be connected in accordance with randomization group. The day after the procedure, a chest x-ray, EKG and pacemaker evaluation will be performed. An echocardiogram will be obtained at 3 months post procedure. At 6 and 12 months post procedure, EKG rhythm strips will be obtained from patients' standard of care remote pacemaker monitoring systems.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years old.
2. With signed consent.
3. Pacemaker indication according to 2018 American College of Cardiology/American Heart Association/Heart Rhythm Society Guideline on the Evaluation and Management of Patients with Bradycardia and Cardiac Conduction Delay. With one or both of the following:

   1. Symptomatic sinus node dysfunction.
   2. Symptomatic Atrioventricular (AV) block or high degree AV block.
   3. Tachy-Brady syndrome

Exclusion Criteria:

1. Previously implanted cardiac pacing devices except transvenous temporary pacemaker.
2. Patients who are eligible for appropriate cardiac resynchronization therapy(CRT) or implantable cardiovert defibrillator (ICD) implantation
3. Patients with prior septal myectomy
4. Patients with prior surgical or transcatheter aortic valve replacement
5. Anatomy precluding implant evaluated during the screening or identified during the procedure.
6. Those without ability to achieve selective His bundle pacing evaluated during the screening or identified during the procedure
7. Pregnant women

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Haines, MD, Principal Investigator — Beaumont
Locations (2):
- United States (2):
  - Beaumont Health System, Royal Oak, Michigan
  - Beaumont Health System, Troy, Michigan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: 3 Month Follow up
Arm/Group | Selective or Non Selective His Bundle Pacing | Left Bundle Area Pacing
Started | 3 | 6
Completed | 3 | 5
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1
Period: 6month Follow up
Arm/Group | Selective or Non Selective His Bundle Pacing | Left Bundle Area Pacing
Started | 3 | 5
Completed | 2 | 2
Not Completed | 1 | 3
Not completed — Physician Decision | 1 | 3
Period: 12 Month Follow up
Arm/Group | Selective or Non Selective His Bundle Pacing | Left Bundle Area Pacing
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Selective or Non Selective His Bundle Pacing | Left Bundle Area Pacing | Total
Number analyzed (Participants) | 3 | 6 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.67 (9.02) | 78.83 (9.7) | 79.44 (8.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 2 | 4 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Ventricular Capture Threshold, 3 Months Unipolar or Bipolar
Description: Ventricular capture threshold is the minimum amplitude of electrical signal from the pacemaker that consistently results in capture of the ventricular myocardium (normal contraction of the ventricle after electrical depolarization) with a 1.0 millisecond pulse width setting in unipolar or Bipolar output modes, measured in volts. During pacemaker placement, the ideal ventricular capture threshold is determined by delivering a series of pulses starting at 0.75 volts and increasing by 0.125 V with each trial until consistent ventricular contraction is achieved. Pacemaker settings are programmed using the ventricular capture threshold, adjusted to include a safety margin, and may be re-adjusted over time if clinically necessary. The measurement is automatically recorded within the pacemaker and will be interrogated from the pacemaker device at 3 months post implantation.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: volts
Arm/Group | Selective or Non Selective His Bundle Pacing | Left Bundle Area Pacing
Number analyzed (Participants) | 3 | 5
volts | 0.66 (0.14) | 0.65 (0.13)

2. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF) - Intrinsic Conduction
Description: Percentage of blood pumped from the left ventricle of the heart at each beat with no pacing applied
Time Frame: at index procedure prior to lead fixation
Population: Echocardiogram data not collected for any subject for any outcome in this study.
Arm/Group | Selective or Non Selective His Bundle Pacing | Left Bundle Area Pacing
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Stroke Volume - Intrinsic Conduction
Description: Volume of blood in milliliters pumped from the left ventricle of the heart at each beat with no pacing applied
Time Frame: at index procedure prior to lead fixation
Population: Echocardiogram data not collected for any subject for any outcome in this study
Arm/Group | Selective or Non Selective His Bundle Pacing | Left Bundle Area Pacing
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Mechanical Dyssynchrony of Anterior Left Ventricle Myocardial Wall- Intrinsic Conduction
Description: Time to peak systolic velocity of the anterior left ventricle myocardial wall in milliseconds with no pacing applied, elicited by tissue Doppler
Time Frame: at index procedure prior to lead fixation
Population: Echocardiogram data not collected for any subject for any outcome in this study
Arm/Group | Selective or Non Selective His Bundle Pacing | Left Bundle Area Pacing
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Mechanical Dyssynchrony of Inferior Left Ventricle Myocardial Wall- Intrinsic Conduction
Description: Time to peak systolic velocity of the inferior left ventricle myocardial wall in milliseconds with no pacing applied, elicited by tissue Doppler
Time Frame: at index procedure prior to lead fixation
Population: Echocardiogram data not collected for any subject for any outcome in this study
Arm/Group | Selective or Non Selective His Bundle Pacing | Left Bundle Area Pacing
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Mechanical Dyssynchrony of Inferior-septal Left Ventricle Myocardial Wall- Intrinsic Conduction
Description: Time to peak systolic velocity of the inferior-septal left ventricle myocardial wall in milliseconds with no pacing applied, elicited by tissue Doppler
Time Frame: at index procedure prior to lead fixation
Population: Echocardiogram data not collected for any subject for any outcome in this study
Arm/Group | Selective or Non Selective His Bundle Pacing | Left Bundle Area Pacing
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Mechanical Dyssynchrony of Left Ventricle Anterior-septal Myocardial Wall- Intrinsic Conduction
Description: Time to peak systolic velocity of the left ventricle anterior-septal myocardial wall in milliseconds with no pacing applied, elicited by tissue Doppler
Time Frame: at index procedure prior to lead fixation
Population: Echocardiogram data not collected for any subject for any outcome in this study
Arm/Group | Selective or Non Selective His Bundle Pacing | Left Bundle Area Pacing
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Mechanical Dyssynchrony of Lateral Left Ventricle Myocardial Wall- Intrinsic Conduction
Description: Time to peak systolic velocity of the lateral left ventricle myocardial wall in milliseconds with no pacing applied, elicited by tissue Doppler
Time Frame: at index procedure prior to lead fixation
Population: Echocardiogram data not collected for any subject for any outcome in this study
Arm/Group | Selective or Non Selective His Bundle Pacing | Left Bundle Area Pacing
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Mechanical Dyssynchrony of Inferior-lateral Left Ventricle Myocardial Wall- Intrinsic Conduction
Description: Time to peak systolic velocity of the inferior-lateral left ventricle myocardial wall in milliseconds with no pacing applied, elicited by tissue Doppler
Time Frame: at index procedure prior to lead fixation
Population: Echocardiogram data not collected for any subject for any outcome in this study
Arm/Group | Selective or Non Selective His Bundle Pacing | Left Bundle Area Pacing
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: QRS Duration - Intrinsic Conduction
Description: Duration (time in milliseconds) of the QRS wave complex interval measured from the end of the PR interval to the end of the S wave measured on a 12-lead electrocardiogram, with intrinsic conduction (prior to implantation of the pacemaker), indicating the length of time required for the electrical depolarization of the right and left ventricles of the heart and contraction of the large ventricular muscles.
Time Frame: at index procedure prior to lead fixation
Population: One patient in HIS bundle pacing group had no data for this outcome.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Selective or Non Selective His Bundle Pacing | Left Bundle Area Pacing
Number analyzed (Participants) | 2 | 6
milliseconds | 145 (21.21) | 124.83 (26.63)

11. Secondary Outcome: QRS Duration After Lead Fixation
Description: Duration (time in milliseconds) of the QRS wave complex interval measured from the end of the PR interval to the end of the S wave measured on a 12-lead electrocardiogram, with intrinsic conduction (prior to implantation of the pacemaker), indicating the length of time required for the electrical depolarization of the right and left ventricles of the heart and contraction of the large ventricular muscles. A normal duration is between 80-100 milliseconds. A QRS duration of greater than 120 milliseconds is considered abnormal.
Time Frame: at index procedure following final lead fixation
Population: One patient in left bundle area pacing group had missing data for this outcome
Measure: Mean (Standard Deviation); unit: millliseconds
Arm/Group | Selective or Non Selective His Bundle Pacing | Left Bundle Area Pacing
Number analyzed (Participants) | 3 | 5
millliseconds | 129.33 (35.8) | 129.8 (10.83)

12. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF) - 3 Months
Description: LVEF is the percentage of blood pumped from the left ventricle of the heart with each beat. It is calculated as the fraction of chamber volume ejected in systole (stroke volume) in relation to the volume of the blood in the ventricle at the end of diastole (end-diastolic volume). Volumes are measured via ultrasound in an echocardiogram. A healthy LVEF ranges from 50-70%. LVEF less than 40% are considered low and indicate some degree of heart failure. LVEF less than 35% are considered dangerous and indicate a subject at risk for arrhythmia.
Time Frame: 3 months
Population: Echocardiogram data not collected for any subject for any outcome in this study
Arm/Group | Selective or Non Selective His Bundle Pacing | Left Bundle Area Pacing
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Stroke Volume - 3 Months
Description: Volume of blood in milliliters pumped from the left ventricle of the heart at each beat 3 months after final pacing lead fixation
Time Frame: 3 months
Population: Echocardiogram data not collected for any subject for any outcome in this study
Arm/Group | Selective or Non Selective His Bundle Pacing | Left Bundle Area Pacing
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Mechanical Dyssynchrony of Anterior Left Ventricle Myocardial Wall - 3 Months
Description: Time to peak systolic velocity of the anterior left ventricle myocardial wall in milliseconds 3 months after final pacing lead fixation, elicited by tissue Doppler
Time Frame: 3 months
Population: Echocardiogram data not collected for any subject for any outcome in this study
Arm/Group | Selective or Non Selective His Bundle Pacing | Left Bundle Area Pacing
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Mechanical Dyssynchrony of Inferior Left Ventricle Myocardial Wall - 3 Months
Description: Time to peak systolic velocity of the inferior left ventricle myocardial wall in milliseconds 3 months after final pacing lead fixation, elicited by tissue Doppler
Time Frame: 3 months
Population: Echocardiogram data not collected for any subject for any outcome in this study
Arm/Group | Selective or Non Selective His Bundle Pacing | Left Bundle Area Pacing
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Mechanical Dyssynchrony of Left Ventricle Anterior-septal Myocardial Wall - 3 Months
Description: Time to peak systolic velocity of the left ventricle anterior-septal myocardial wall in milliseconds 3 months after final pacing lead fixation, elicited by tissue Doppler
Time Frame: 3 months
Population: Echocardiogram data not collected for any subject for any outcome in this study
Arm/Group | Selective or Non Selective His Bundle Pacing | Left Bundle Area Pacing
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Mechanical Dyssynchrony of Left Ventricle Inferior-septal Myocardial Wall- 3 Months
Description: Time to peak systolic velocity of the left ventricle inferior-septal myocardial wall in milliseconds 3 months after final pacing lead fixation, elicited by tissue Doppler
Time Frame: 3 months
Population: Echocardiogram data not collected for any subject for any outcome in this study
Arm/Group | Selective or Non Selective His Bundle Pacing | Left Bundle Area Pacing
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Mechanical Dyssynchrony of Lateral Left Ventricle Myocardial Wall- 3 Months
Description: Time to peak systolic velocity of the lateral left ventricle myocardial wall in milliseconds 3 months after final lead fixation, elicited by tissue Doppler
Time Frame: 3 months
Population: Echocardiogram data not collected for any subject for any outcome in this study
Arm/Group | Selective or Non Selective His Bundle Pacing | Left Bundle Area Pacing
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Mechanical Dyssynchrony of Inferior-lateral Left Ventricle Myocardial Wall- 3 Months
Description: Time to peak systolic velocity of the inferior-lateral left ventricle myocardial wall in milliseconds 3 months after final lead fixation, elicited by tissue Doppler
Time Frame: 3 months
Population: Echocardiogram data not collected for any subject for any outcome in this study
Arm/Group | Selective or Non Selective His Bundle Pacing | Left Bundle Area Pacing
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: QRS Duration- 3 Months
Description: Duration (time in milliseconds) of the QRS wave complex interval measured from the end of the PR interval to the end of the S wave measured on a 12-lead electrocardiogram, 3 months after final pacing lead fixation, indicating the length of time required for the electrical depolarization of the right and left ventricles of the heart and contraction of the large ventricular muscles. A normal duration is between 80-100 milliseconds. A QRS duration of greater than 120 milliseconds is considered abnormal.
Time Frame: 3 months
Population: 1 patient in the left bundle area pacing group had data missing for this outcome
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Selective or Non Selective His Bundle Pacing | Left Bundle Area Pacing
Number analyzed (Participants) | 3 | 4
milliseconds | 108.67 (19.22) | 123 (46.26)

21. Secondary Outcome: Capture Threshold - 6 Months, Unipolar or Bipolar
Description: Ventricular capture threshold is the minimum amplitude of electrical signal from the pacemaker that consistently results in capture of the ventricular myocardium (normal contraction of the ventricle after electrical depolarization) with a 1.0 millisecond pulse width setting in unipolar or Bipolar output modes, whichever value is lower, measured in volts. During pacemaker placement, the ideal ventricular capture threshold is determined by delivering a series of pulses starting at 0.75 volts and increasing by 0.125 V with each trial until consistent ventricular contraction is achieved. Pacemaker settings are programmed using the ventricular capture threshold, adjusted to include a safety margin, and may be re-adjusted over time if clinically necessary. The measurement is automatically recorded within the pacemaker and will be interrogated from the pacemaker device at 3 months post implantation.
Time Frame: 6 months
Population: 4 patients completed data collection for 6 month follow-up
Measure: Mean (Standard Deviation); unit: Volts
Arm/Group | Selective or Non Selective His Bundle Pacing | Left Bundle Area Pacing
Number analyzed (Participants) | 2 | 2
Volts | 1.18 (0.79) | 0.93 (0.08)

22. Secondary Outcome: Capture Threshold - 12 Months, Unipolar or Bipolar
Description: as for outcome 21
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Volts
Arm/Group | Selective or Non Selective His Bundle Pacing | Left Bundle Area Pacing
Number analyzed (Participants) | 2 | 2
Volts | 1.31 (0.61) | 1.12 (0)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Selective or Non Selective His Bundle Pacing | Left Bundle Area Pacing
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/6
Other Adverse Events (participants affected / at risk) | 0/3 | 0/6

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects and ECHO data not available for any subject.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-23): https://cdn.clinicaltrials.gov/large-docs/14/NCT04093414/Prot_SAP_000.pdf